CLINICAL TRIAL: NCT03817632
Title: Prospective, Multicenter, Observational, Comparative Clinical Trial on the Equivalence of Two Different OrthoPilot® Navigation System Generations Applied for Computer-assisted Total Knee Arthroplasty
Brief Title: Orthopilot Elite Post-Market Clinical Follow-Up
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1708
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Degenerative Osteoarthritis; Rheumatoid Arthritis; Posttraumatic Arthropathy; Instability, Joint; Stiffness of Knee, Not Elsewhere Classified; Deformity of Knee
Keywords: Navigation; Computer Assisted Orthopedic Surgery; OrthoPilot®; Total Knee Arthroplasty
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid; Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A Standard: Computer assisted primary total knee replacement with OrthoPilot FS 101 navigation system and Software 5.1
  Interventions: Device: Computer assisted primary total knee replacement with OrthoPilot FS101 navigation system and Software 5.1
- B Elite: Computer assisted primary total knee replacement with OrthoPilot Elite navigation system and Software 6.0
  Interventions: Device: Computer assisted primary total knee replacement with OrthoPilot Elite navigation system and Software 6.0

INTERVENTIONS:
Device: Computer assisted primary total knee replacement with OrthoPilot FS101 navigation system and Software 5.1 — Computer Assisted Total Knee Replacement with the OrthoPilot FS101 and the software TKA 5.1
  Groups: A Standard
Device: Computer assisted primary total knee replacement with OrthoPilot Elite navigation system and Software 6.0 — Computer Assisted Total Knee Replacement with the with the OrthoPilot Elite and the software TKA 6.0
  Groups: B Elite

SUMMARY:
Prospective, multicenter, observational, comparative clinical trial on the equivalence of two different OrthoPilot® navigation system generations applied for computer-assisted total knee arthroplasty

DETAILED DESCRIPTION:
The study is designed as a prospective, non-interventional, multicenter, comparative cohort study. The product under investigation will be used in routine clinical practice and according to the authorized Instructions for Use (IfU). Those data that are obtained in routine clinical use will be documented in the Case Report Form (CRF).

The study design is based on a two-arms design. The patients for the both groups will be recruited consecutively, starting with group A. The study will prove the equivalence of the groups regarding the outcome of the postoperative lower limb alignment (mechanical leg axis) and any deviation >3° from neutral alignment is defined as an outlier.

ELIGIBILITY:
Inclusion: Inclusion Criteria:

* Patients with indication for Total Knee Arthroplasty using the Aesculap OrthoPilot® navigation system and a corresponding primary implant
* Dated and signed informed consent

Exclusion: Exclusion Criteria

* Pregnancy
* Patients < 18 years
* Patients unable to participate at the follow-up examination (physically, mentally)
* Previous joint replacement at the indexed knee

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Rate of Lower Limb Alignment inside the range of 0±3° | three months postoperatively
  A postoperative lower limb alignment of the knee prosthesis in reference to the mechanical leg axis (3, 18) outside the range of ± 3° is defined as the outlier. The outlier rates will be used as the efficacy criterion for groups comparison

SECONDARY OUTCOMES:
Lower limb alignment of the knee prosthesis in reference to the mechanical leg axis | 3 months postoperatively
  The outcome and function of a prosthesis is influenced by the postoperative alignment of the leg and the orientation in reference to the axis. Incorrect positioning can lead to an increased implant wear and functional limitations (23, 24). The aim of a postoperative alignment within 3° varus to 3° valgus will be assessed using long leg x-rays 3-4 months postoperatively.
Improvement of Knee Society Score (KSS) | preoperatively and three months postoperatively
  The KSS score is composed of two subgroups and has a maximum score of 200.
Improvement of Oxford Knee Score (OKS) | preoperatively and three months postoperatively
  A patient-reported outcome instrument which contains 12 questions on activities of daily living that assess function and residual pain in patients undergoing total knee replacement (TKR) arthroplasty. Oxford Knee Score has a maximum of 48 points indicating satisfactory knee function
Improvement of Quality of Life (EQ-5D-5L) | preoperatively and three months postoperatively
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Learning Curve | Intraoperatively
  The first 10 cases of each surgeon shall be excluded from the main analysis. The results of the first 10 cases ("learning curve") shall be assessed separately and compared with the "10 plus" cases ("routine cases") as a secondary learning curve analysis. The potential learning curve will be assessed measuring the intraoperative surgery time in reference to the already performed procedures of each surgeon
Intraoperative handling of soft- and hardware components | Intraoperatively
  Aim of this study is also to document any upcoming problems or limitations the operating surgeon has with the new components of the OrthoPilot® Elite hardware system and the new software application TKA 6.0 for the implantation of primary total knee endoprosthesis. Intraoperatively documented results of the navigation system will be recorded and integrated into the final analysis. Potential problems or comments will be analysed descriptively.
(Serious) Adverse Device Effects | up to 3 months postoperatively
  As part of the follow-up examination, any upcoming (serious) adverse device events or effects related or not related to the product under investigation, will be documented in the dedicated Case Report Forms. Recorded complications will be categorized and analyzed in order to assess the safety of the OrthoPilot® navigation system

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Uniklinikum Freiburg, Freiburg im Breisgau
  - Schönkliniken Klinikum Eilbek, Hamburg